CLINICAL TRIAL: NCT05239572
Title: Scaling Up Non-Communicable Diseases Interventions in South East Asia
Brief Title: Scaling Up NCD Interventions in South East Asia
Acronym: SUNI-SEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: University of Groningen (Other); University of Passau (Unknown); Universitas Sebelas Maret (Other); Health Strategy and Policy Institute (Unknown); Trnavska Universita v Trnava (Unknown); HelpAge International (Unknown); Thai Nguyễn University of Medicine and Pharmacy (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 202100908
Record Dates: First submitted 2022-01-03; First posted 2022-02-15 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension; Cardiovascular Diseases
Keywords: prevention; early diagnosis; lifestyle intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Cardiovascular Diseases; Disease | interventions — Mass Screening; Counseling; Risk Factors; Therapeutics

STUDY DESIGN:
Intervention Model Description: In Vietnam members from 60 Intergenerational Self Help Clubs have been screened for diabetes and cardiovascular diseases. (total 5,000 persons) In Myanmar members from 15 Intergenerational Solidarity Groups have undergone screening for diabetes and cardiovascular diseases using an internet application. (total 1850 persons) In Indonesia, visitors of 20 Posbindu programmes were offered screened for diabetes and hypertension in Central and East Java (10,000 persons)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening and early detection of diabetes and cardiovascular diseases (Experimental): Screening for NCDs based on questionnaire concerning vital information, lifestyle, simple measures of length, bodyweight, BMI, blood pressure, application of FinRisk score and WHO risk score.
  Health promotion and lifestyle counselling and referral to PHC facilities for further diagnosis and treatment.
  Interventions: Combination Product: screening, prevention and counselling

INTERVENTIONS:
Combination Product: screening, prevention and counselling — Screening in Intergenerational solidarity clubs in Myanmar and Vietnam and in Posbindu programme in Indonesia
  Other Names: lifestyle coaching for persons with risk factors for NCDs; referral to primary healthcare facilities for further diagnosis and treatment; simple treatment of NCDs at primary healthcare level; Online monitoring and counselling for risk factors for NCDs

SUMMARY:
The SUNI-SEA study is an intervention study that measures effectiveness and cost-effectiveness of prevention and early diagnosis of diabetes and cardiovascular diseases in communities and primary healthcare (PHC) facilities in Indonesia, Myanmar and Vietnam.

DETAILED DESCRIPTION:
The study takes place in Vietnam and Indonesia in Intergenerational Self-Help Clubs (ISHGs), where community members assemble for activities concerning social, economical improvement and health and well-being. Volunteers in these ISHGs are trained in performing screening for diabetes and cardiovascular diseases and counselling participants concerning healthy living, or referral to primary healthcare facilities, if needed. At PHC level further diagnosis and if needed treatment is provided and referral back to ISHGs is done for lifestyle interventions.

In Indonesia screening takes place in the Posbindu programme, where trained volunteers (cadres) screen and counsel participants. If needed referral to Puskesmas (primary healthcare facilities is done, where further diagnosis and treatment takes place. Activities for health promotion and lifestyle interventions take place under supervision of the Posbindu programme.

In Myanmar and Indonesia individual monitoring and health education of participants is done through mobile applications.

Measuring of uptake, follow-up and adherence to interventions is done through routine data collection, through surveys, and through semi-structured interviews and focus group discussions.

ELIGIBILITY:
Inclusion Criteria:

* All adults living in geographical area where research takes place

Exclusion Criteria:

* Persons who are not able to come to location of screening, due to illness or other chronic condition causing immobility.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16850 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Uptake of NCD screening offered in communities | 18 months from offering screening options in communities until measuring uptake
  Number of adults eligible for NCD screening in communities who participate in screening
Adherence to follow-up advice | 12 months from counselling and advice to individual until measuring adherence to follow-up that has been recommended
  Percentage of participants in screening who follow up on recommendations given during screening (referral, lifestyle change)
Uptake of health education (health promotion, awareness of risk factors) | 12 year between first health education session and measuring uptake (based on participants' lists)
  Percentage of adults above 21 years in communities participating in one or more health education sessions offered

SECONDARY OUTCOMES:
Unit costs of screening, prevention and early diagnosis of NCDs per Quality Adjusted Life Year gained | 18 months between starting calculation of costs of interventions and assessment of final assessment of benefits
  Unit costs of NCD screening, prevention, early diagnosis intervention per Quality Adjusted Life Year gained
Cost-effectiveness of NCD interventions | 18 months between baseline survey and endline survey
  Comparison of costs and effects between intervention and business as usual, using diff in diff method

OTHER OUTCOMES:
Impact of training of community health volunteers in NCD interventions on knowledge attitudes and practices of volunteers | 6 months between provision of training to community health volunteers and measuring their skills, knowledge and attitudes
  Difference in knowledge, attitudes and practices (KAP) of volunteers in ISHCs in Myanmar and Vietnam, and cadres in Posbindu in Indonesia as result of training offered in the research project, measured by pre- and post-training KAP survey and six months after training.
Impact of training of community health volunteers on their performance in NCD interventions. | 6 months between provision of training to community health volunteers and measuring their performance
  Performance of community health volunteers six months after training, measured by observational study, with measuring adherence to standard operating procedures for screening for NCDs and health education.

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Postma, PhD, Principal Investigator — University Medical Center Groningen; Robert Lensink, PhD, Principal Investigator — University of Groningen; Ari Probandari, PhD, Principal Investigator — University Sebelas Maret; Giang Nguyen Hoang, MPH, Principal Investigator — Health Strategy and Policy Institute; Anil Kumar Indira Krishna, PhD, Principal Investigator — HelpAge International; Michael Grimm, PhD, Principal Investigator — University of Passau
Locations (1):
- Health Strategy and Policy Institute, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Following open research guidelines of European Union data will be shared about screening, follow-up and referral. Data collected in cos-effectiveness analysis will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available after July 2023 and will be available for period according to regulations of European Union
Access Criteria: On request for researchers performing secondary data analysis
URL: http://www.suni-sea.org

REFERENCES:
- [Derived] Hanifa RS, Rokhman MR, Fritz M, Widyaningsih V, Febrinasari RP, Koot JAR, Postma MJ, van der Schans J. Cost-effectiveness of community-based type 2 diabetes prevention and control in Indonesia: a health economics modelling study. BMJ Public Health. 2025 Oct 7;3(2):e002161. doi: 10.1136/bmjph-2024-002161. eCollection 2025. PMID 41069974
- [Derived] Fritz M, Grimm M, My Hanh HT, Koot JAR, Nguyen GH, Nguyen TP, Probandari A, Widyaningsih V, Lensink R. Effectiveness of community-based diabetes and hypertension prevention and management programmes in Indonesia and Viet Nam: a quasi-experimental study. BMJ Glob Health. 2024 May 22;9(5):e015053. doi: 10.1136/bmjgh-2024-015053. PMID 38777393
- See also: dedicated research project website — http://www.suni-sea.org